CLINICAL TRIAL: NCT05199350
Title: Distinguishing Participant Groups Using Autonomic Dysfunction
Status: Completed | Type: Observational
Sponsor: DyAnsys, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CS013
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-08

CONDITIONS: Diabetes
Keywords: Impaired Fasting Glucose; Autonomic Dysfunction Measurement; Heart Rate Variability; Vital Signs Monitoring
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Population including people with NGT, IFG and IGT and diabetes.: Normal Glucose Tolerance (NGT) is defined as a plasma glucose concentration i.e < 140 mg/dl.
  IFG is defined by an elevated fasting plasma glucose (FPG) concentration i.e ≥ 100 and < 126 mg/dl.
  IGT is defined by an elevated post-prandial plasma glucose concentration i.e ≥140 and < 200 mg/dl.
  Presence of confirmed diabetes (HbA1c level > 6.4 %) without complications i.e no neuropathy, no retinopathy, no nephropathy etc.
  Presence of confirmed diabetes (HbA1c level > 6.4 %) with at least one of the above complications.
  Interventions: Other: Device Name: ANSiscope

INTERVENTIONS:
Other: Device Name: ANSiscope — Heart rate variability measurement and vital signs monitoring will be performed on all subjects.

SUMMARY:
A study population with impaired fasting glucose levels, impaired glucose tolerance levels and diabetes (with or without complications) along with healthy patients will be chosen as participants. Their vital signs and their ECG (electrocardiograph) will be recorded during their only visit. Data analysis will be performed using the vital signs parameters. The RR intervals from the ECG will be analyzed by 5 different techniques to determine the best technique that stratifies the subjects the most accurately.

DETAILED DESCRIPTION:
The Autonomic Nervous System (ANS) is a fundamental part of the nervous system in the body. And yet, there is no technique to test or measure the health and functioning of a person's autonomic nervous system.This type of study will determine the most accurate methodology to test the autonomic nervous system through heart rate variability (HRV) monitoring and gain vital information to distinguish patient groups in the diabetic population.

There is no gold standard for measuring autonomic dysfunction. Currently the method of power spectral analysis is finding very wide usage. It Is known that power spectral analysis does not discriminate the two subsystems of the ANS well. There are other beat to beat methodologies that have not yet gained traction. The reason for conducting this trial is to take a group of subjects in various stages of impaired fasting glucose, impaired glucose tolerance and diabetes (with and without complications) and determine which methodology stratifies these subjects most accurately.

Our study aims to introduce a new measurement method named the 'Beat to Beat' (BB) method for gauging autonomic dysfunction in patients. The investigators hope to observe that the average beat to beat method (BB) score could help discriminating diabetic patients into the following five distinct groups from the pilot study:

1. Normal Glucose Tolerance (NGT) is defined as a plasma glucose concentration i.e < 140 mg/dl.
2. Impaired Fasting Glucose (IFG) is defined by an elevated fasting plasma glucose (FPG) concentration i.e ≥ 100 and < 126 mg/dl.
3. Impaired Glucose Tolerance (IGT) is defined by an elevated post-prandial plasma glucose concentration i.e ≥140 and < 200 mg/dl.
4. Presence of confirmed diabetes (HbA1c level > 6.4 %) without complications i.e no neuropathy, no retinopathy, no nephropathy etc.
5. Presence of confirmed diabetes (HbA1c level > 6.4 %) with at least one of the above complications.

By showing that this measurement bears no relationship to the other four vital signs parameters (heart rate, blood oxygenation, blood pressure, body temperature), it will prove the necessity of this measurement in addition to the four vital signs for distinguishing patient groups among the diabetic population.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent
2. Age between 18 to 85
3. Body Mass Index (BMI) between 25 and 40 kg/m2
4. Individuals with normal glucose levels, pre-diabetes and diabetes Type 2 for at least 1 year (diagnosed by ADA criteria) and up to 20 years
5. Stable dose of meds for 3 months
6. Stable diet and lifestyle for 3 months
7. Medical history without clinically significant abnormalities

Exclusion Criteria:

1. Have a disorder that would impede performing the HRV measurement procedure (i.e., abnormal cardiac rhythm, heart disease, including coronary artery disease, angina, and arrhythmia, cardiac pacemaker, stroke, panic attack, cognitive impairment, renal failure)
2. Chronic disease (e.g. HIV, Cushing syndrome, CKD, acromegaly, active hyperthyroidism etc.)
3. Cancer and anticancer treatment in the last 5 years
4. Pregnancy or lactation
5. Subjects with major physical disability
6. Subjects with previous history of cerebrovascular accident
7. Any disorder, which in the investigator's opinion might jeo

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults of either sex with various stages of impaired fasting glucose tolerance levels and diabetes (with or without complications) will be considered as study population.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Determination of autonomic dysfunction by subject | The measurement will happen in a single visit i.e 1 day.
  The ANSiScope Plus will be used to determine the BB (beat to beat) score through heart rate variability measurements.

SECONDARY OUTCOMES:
Establish the absence of any relationship of autonomic dysfunction (AD) to any other vital signs parameters. | The measurement will happen in a single visit i.e 1 day.
  Investigate the importance of measuring the autonomic dysfunction in the presence of other vital signs measurements (heart rate, body temperature, blood oxygenation and blood pressure)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mathangi Dr D.C, Prof &Head M.SC., Phd, Principal Investigator — Sri Rachandra Institute of HigherEducation And Research hospital; priscilla Dr johnson, MBBS,MD, DNB, PhD, Study Chair — Sri Rachandra Institute of HigherEducation And Research hospital; shriram Dr Mahadevan, Principal Investigator — Sri Rachandra Institute of HigherEducation And Research hospital; Divyalakshmi Dr Divyalakshmi k, MBBS,MD, Study Director — Sri Rachandra Institute of HigherEducation And Research hospital
Locations (1):
- Sri Rachandra Institute of HigherEducation And Research, Chennai, Tamil Nadu, India